CLINICAL TRIAL: NCT01406418
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled Study in Healthy Subjects to Assess the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of CR6261, a Monoclonal Antibody Against Influenza A Viruses, Following Single-Dose Intravenous Administration
Brief Title: Assessment of CR6261, a Monoclonal Antibody Against the Influenza A Virus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Crucell Holland BV (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FLU-M6-C001; DMID Protocol 11-0025 (Other Grant/Funding Number: DMID HHSN272200900060C)
Record Dates: First submitted 2011-07-28; First posted 2011-08-01 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Influenza
Keywords: Influenza; Virus; Monoclonal; Antibody; Immunization; Treatment
MeSH Terms: conditions — Influenza, Human; Virus Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (12):
- Cohort 1: CR6261 (Experimental): 2 mg/kg CR6261
  Interventions: Biological: CR6261 2 mg/kg
- Cohort 1: Placebo (Placebo Comparator): 5% dextrose in water
  Interventions: Biological: Placebo
- Cohort 2: CR6261 (Experimental): 5 mg/kg CR6261
  Interventions: Biological: CR6261 5 mg/kg
- Cohort 2: Placebo (Placebo Comparator): 5% dextrose in water
  Interventions: Biological: Placebo
- Cohort 3: CR6261 (Experimental): 15 mg/kg CR6261
  Interventions: Biological: CR6261 15 mg/kg
- Cohort 3: Placebo (Placebo Comparator): 5% dextrose in water
  Interventions: Biological: Placebo
- Cohort 4: CR6261 (Experimental): 30 mg/kg CR6261
  Interventions: Biological: CR6261 30 mg/kg
- Cohort 4: Placebo (Placebo Comparator): 5% dextrose in water
  Interventions: Biological: Placebo
- Cohort 5: CR6261 (Experimental): 50 mg/kg CR6261
  Interventions: Biological: CR6261 50 mg/kg
- Cohort 5: Placebo (Placebo Comparator): 5% dextrose in water
  Interventions: Biological: Placebo
- Cohort 6: CR6261 (Experimental): 30 mg/kg CR6261
  Interventions: Biological: CR6261 30 mg/kg
- Cohort 6 Placebo (Placebo Comparator): 5% dextrose in water
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CR6261 2 mg/kg — Administered as a single 2-hour intravenous infusion
  Arms: Cohort 1: CR6261
Biological: CR6261 5 mg/kg — Administered as a single 2-hour intravenous infusion
  Arms: Cohort 2: CR6261
Biological: CR6261 15 mg/kg — Administered as a single 2-hour intravenous infusion
  Arms: Cohort 3: CR6261
Biological: CR6261 30 mg/kg — Administered as a single 2-hour intravenous infusion
  Arms: Cohort 4: CR6261; Cohort 6: CR6261
Biological: CR6261 50 mg/kg — Administered as a single 2-hour intravenous infusion
  Arms: Cohort 5: CR6261
Biological: Placebo — Administered as a single 2-hour intravenous infusion
  Arms: Cohort 1: Placebo; Cohort 2: Placebo; Cohort 3: Placebo; Cohort 4: Placebo; Cohort 5: Placebo; Cohort 6 Placebo

SUMMARY:
The purpose of this study is to assess in healthy subjects the safety, tolerability, pharmacokinetics and immunogenicity of single escalating doses of CR6261, a monoclonal antibody against influenza A viruses.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled dose escalation study will enroll up to 6 cohorts of healthy subjects. Eight subjects will be enrolled in each cohort (1 to 5) and will receive a single 2-hour intravenous infusion of CR6261 (6 subjects) or placebo (2 subjects) on Day 1. Subjects will be dosed in pairs of two. Once all subjects in a cohort have completed Study Day 8, the preliminary safety data will be reviewed. Provided that no safety issues are identified, dose escalation to the subsequent cohort may be permitted.

To obtain additional data at the 30 mg/kg dose level, a sixth cohort will be enrolled after the preliminary safety and tolerability of the 30 mg/kg dose in Cohort 4 is demonstrated. Cohort 6 will be comprised of 24 subjects (randomized 5 : 1 to CR6261 or placebo) following the same visit schedule as subjects in Cohorts 1-5.

ELIGIBILITY:
INCLUSION CRITERIA

1. Adult male and female subjects aged 18 to 50 years on Study Day 1.
2. Body mass index between 18 and 30 (kg/m2) by nomogram or calculation; body weight between 50 kg and 100 kg.
3. Has acceptable blood pressure and heart rate parameters within the normal limits (systolic = 88-140 mmHg; diastolic = 50 to <90 mmHg; heart rate = 46 to 100 bpm).
4. Healthy as determined by pre-study medical history, physical examination, and laboratory assessments.
5. Able and willing to give written informed consent.
6. Has the ability to complete the follow-up period of 75 days as required by the protocol.
7. Subjects must agree to abstain from alcohol intake 24 hours before administration of study drug, during the inpatient period of the study and 24 hours prior to all other outpatient clinic visits.
8. Subjects must agree to not use OTC medications (including aspirin, decongestants, antihistamines and other NSAIDs), and herbal medication (including, but not limited to, herbal tea, St. John's Wort), within 14 days prior to study drug administration through the final follow-up visit, unless approved by the investigator and medical monitor. Occasional use of acetaminophen/paracetamol at recommended doses (≤ 1 gram/6 hours and ≤ 4 grams/day) and continued pre-existing use of vitamins or multivitamins at recommended doses is allowed.
9. Female subjects must:

   * Be surgically sterile (have had a hysterectomy or bilateral oophorectomy, tubal ligation, or otherwise be incapable of pregnancy), or
   * If heterosexually active, use two effective methods of birth control, including hormonal prescription oral contraceptives, contraceptive injections, contraceptive patch, contraceptive ring, intrauterine device, barrier method (e.g. condoms, diaphragm, or cervical cap), or spermicidal foam, cream, or gel), or
   * Confirm male partner sterilization, or
   * Not be heterosexually active Note: women who are not heterosexually active at screening must agree to utilize two effective methods of birth control if they become heterosexually active during their participation in the study.

   Women must agree to continue using these methods of contraception throughout the study.
10. Females must have a negative urine pregnancy test at both screening and baseline.
11. If a man who is able to father a child and sexually active with a female of childbearing potential, he must agree to use a double barrier method of birth control (e.g. condom with spermicidal foam, cream, or gel) and to not donate sperm during the study.
12. Subjects must agree to avoid strenuous exercise (e.g. long distance running >5 km/day, weight lifting, or any physical activity to which the subject is not accustomed) while confined to the Clinical Unit and for at least 72 hours prior to study drug administration and follow up visits.

EXCLUSION CRITERIA

1. Acute illness at the time of entry into the study (Study Day 1).
2. Temperature >99.5oF (37.5oC) at randomization.
3. Presence of a significant infection or known inflammatory process during screening or at the time of randomization.
4. Presence of acute gastrointestinal symptoms during screening or at the time of randomization (e.g. nausea, vomiting, diarrhea, or heartburn).
5. A diagnosis of influenza infection or any constellation of clinical symptoms consistent with influenza infection (e.g. fever, myalgias, headache, fatigue, non-productive cough, sore throat, and/or rhinorrhea) within 14 days prior to Study Day 1.
6. Received any live virus or bacterial vaccinations within 3 months prior to screening or are expected to receive any live virus or bacterial vaccinations during the study.
7. Received inactivated influenza vaccines within 2 weeks of Study Day 1 or are expected to receive an inactivated influenza vaccine during the study.
8. Any chronic condition requiring prescription or over-the-counter medicine, with the exception of vitamins.
9. Chronic (longer than 14 days) administration of immunosuppressants or other immune modifying drugs within 6 months before administration of the investigational product; oral corticosteroids in dosages of < 0.5 mg/kg/d prednisolone or equivalent and inhaled/nasally/topically administered corticosteroids are permitted.
10. Antibiotic therapy within 7 days before Study Day 1.
11. History and/or presence of any clinically significant disease or disorder such as cardiovascular, pulmonary, renal, hepatic, neurological, gastrointestinal and psychiatric/mental disease/disorders, which, in the opinion of the Principal Investigator may either put the subject at risk because of participation in the study, influence the results of the study or the subject's ability to participate in the study.
12. Previous medical history that may compromise the safety of the subject in the study.
13. Positive serology for the human immunodeficiency virus (HIV) 1 or 2 antibody, hepatitis C virus antibody or hepatitis B surface antigen.
14. History of a previous severe allergic reaction with generalized urticaria, angioedema, or anaphylaxis.
15. Known or suspected hypersensitivity to any CR6261 excipients (Sucrose, L-Histidine L-Histidine Monohydrochloride, Polysorbate 20).
16. A history of alcohol or drug abuse within the past 2 years as according to DSM IV.
17. Positive urine test for illicit drugs (opiates, cocaine, amphetamines) during screening and admission (Day -1).
18. Subjects who report current tobacco use of more than 10 cigarettes or 2 cigars per day at screening or anticipate use exceeding this amount at any time during the study.
19. Receipt of any other investigational product within 1 month or 5 half-lives (whichever is longer) before administration of the study investigational product.
20. Participation in any clinical study involving receipt of investigational product, blood or blood products, or donation of blood throughout the duration of the study.
21. Received antibody or biologic therapy (e.g. Ig products, mAbs, or antibody fragments).
22. Subjects who have donated and/or received any blood or blood products within 3 months before administration of the study investigational product or planned donation/receipt throughout the course of the study.
23. Subjects who cannot communicate reliably with the investigator.
24. Any condition that in the opinion of the investigator would complicate or compromise the study, or the well being of the subject.
25. Employee at the clinic, or spouse/relative of the investigator or employees.
26. Has experienced an anaphylactic reaction to latex.
27. Have currently or a past history of thrombocytopenia or bleeding abnormality.
28. Is unable or unwilling to undergo multiple venipunctures because of poor tolerability or lack of easy access to veins.
29. Female subjects who are breastfeeding.
30. Drinks more than 1200 mL (or 5 cups of 240 mL per cup) of tea/coffee/cocoa/cola or other caffeinated beverage per day more than one day per week in the 2 weeks before screening.
31. ECG findings (Screening or Day-1):

    * QTc interval >450 msec;
    * evidence of second- or third-degree atrioventricular (AV) block;
    * pathological Q-waves (defined as Q-wave >40 msec or depth greater than 0.4 - 0.5 mV);
    * evidence of ventricular pre-excitation;
    * electrocardiographic evidence of complete left bundle branch block, right bundle branch block (RBBB), incomplete LBBB;
    * intraventricular conduction delay with QRS duration >120 msec.
32. Laboratory assessments (Screening or Day -1):

    * Hemoglobin below the lower limit of normal (LLN); a lower limit of 13.6 g/dL in males is acceptable;
    * Platelet count, absolute neutrophil count (ANC), or absolute lymphocyte count below LLN (ANC of 1.3 x 10³/µL is acceptable lower limit for African Americans);
    * White blood cell count above the upper limit of normal (ULN) or below the LLN (3.2 x 10³/µL is acceptable lower limit for African Americans);
    * Creatinine above the ULN;
    * PT or PTT above the ULN;
    * ALT, AST, GGTP, ALP, amylase, lipase, or total bilirubin ≥ 1.1 times the ULN (values below the LLN are not considered clinically significant).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2013-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Adverse events and changes in laboratory parameters and vital signs as measures of safety and tolerability of single escalating doses of CR6261 | From baseline to 75 days post-dose

SECONDARY OUTCOMES:
Assessment of pharmacokinetics of single escalating doses of CR6261 | From baseline to 75 days post-dose
  Pharmacokinetic parameters include area under the serum concentration-time curve from zero to the time of the last measurable concentration (AUC0-t), area under the serum concentration-time curve from zero to infinity (AUC0-inf), maximum concentration (Cmax), time of Cmax (tmax), systemic clearance (CL), terminal elimination half life (t1/2), etc.
Assessment of antibodies binding to CR6261 as a measure of immunogenicity of single escalating doses of CR6261 | From baseline to 75 days post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Lisbon, MD, Principal Investigator — Quintiles, Inc.
Locations (1):
- Quintiles Early Clinical Development, Overland Park, Kansas, United States